CLINICAL TRIAL: NCT03080623
Title: Ultrasound-based Diagnostic Model for Differentiating Malignant Breast Lesion From Benign Lesion
Status: Completed | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Tao OUYANG, Chairman of Breast Center of Beijing Cancer Hospital, Peking University
Other Study IDs: D161100000816006
Record Dates: First submitted 2017-02-24; First posted 2017-03-15 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer Female; Diagnoses Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast biopsy pathology
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspicious breast lesions: women with Suspicious breast lesions, who need to receive breast ultrasound will be collected in this cohort. According to the diagnosis of breast ultrasound，patients will be assigned to breast biopsy or follow-up

SUMMARY:
This study proposed to construct an ultrasound-based diagnostic model for Differentiating Malignant Breast Lesion From Benign Lesion. This study contains both retrospective and prospective part, which are designed for model construction and independent validation, respectively.This study aims to construct an easy-to-use ultrasound-based model, prove the efficacy of the model for identifying malignant breast lesion from benign lesion, and finally promote the application of this diagnostic model in more clinics.

ELIGIBILITY:
Inclusion Criteria:

* female
* with single breast lesion(maximum diameter>0.8 cm)
* agree to receive follow-up in six months and take the second breast ultrasound six month after the first breast ultrasound, if a benign diagnosis is achieved at the first ultrasound
* sign the informed consent

Exclusion Criteria:

* lost to follow-up
* failed to take the second breast ultrasound six month after the first breast ultrasound

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: females with breast lesion who need to receive breast ultrasound to make differential diagnosis of benign and malignant lesion
Sampling Method: Probability Sample
Enrollment: 1981 (Actual)
Dates: Start 2018-09-08 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
breast biopsy proved malignant or benign lesion | between breast ultrasound and biopsy(one week)
  for patients regarded as malignant by the breast ultrasound, breast biopsy results are used as reference test, which determines the breast lesion is malignant or benign
two breast ultrasound identified benign lesion | between first detection of breast lesion and the second ultrasound(six month)
  for patients regarded as benign by the breast ultrasound, they will receive a second breast ultrasound after six month(this is regular examination for patients with first detected breast lesion). If the second ultrasound indicates benign, the lesion will be regarded as benign

CONTACTS AND LOCATIONS:
Overall Officials: Tao Ouyang, Study Chair — Peking University Cancer Hospital & Institute
Locations (4):
- China (4):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Haidian women and children's hospital of beijing, Beijing
  - Shunyi women and children's hospital of Beijing Children's Hospital, Beijing
  - Fourth Hospital of Heibei Medical Hospital, Shijiazhuang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huo L, Tan Y, Wang S, Geng C, Li Y, Ma X, Wang B, He Y, Yao C, Ouyang T. Machine Learning Models to Improve the Differentiation Between Benign and Malignant Breast Lesions on Ultrasound: A Multicenter External Validation Study. Cancer Manag Res. 2021 Apr 16;13:3367-3379. doi: 10.2147/CMAR.S297794. eCollection 2021. PMID 33889025